CLINICAL TRIAL: NCT06299358
Title: The Effect of Foot Massage and Maternal Heart Sound on Colic and Comfort Levels in Infants With Infantile Colic
Brief Title: Interventional Practices and Their Effectiveness in Infants With İnfantyl Colic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Meltem Pepe, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KMU_MPEPE_1
Record Dates: First submitted 2024-01-15; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Nurse's Role; Infantile Colic
Keywords: İnfantyl colic; Neonatal; Pediatric Nurses
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Type and Purpose of the Study The study was designed as a randomized experimental study. Sample of the Study G* Power 3.1.9.7. program was used to calculate the sample size (Faul et al., 2007). As a result of the analysis, the sample size was calculated as 28 people for each of the three groups, and considering the possible data losses, it was decided to take 30 people for each group.
  In the study, computer-aided randomization (random.org) program was used to determine the groups. Stratified randomization was preferred to ensure group similarity. In stratification, the number of weeks of age, gender and feeding patterns of the babies were used. After stratification, block randomization was used to decide which group the babies would be in.
  SPSS 22.0 package program will be used for data analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the study, interviews will be conducted at different times so that mothers or caregivers do not encounter mothers/caregivers in other groups. In this way, participant blinding will be ensured. Since the study will be conducted with newborns, no study will be conducted on other blinding techniques and biases. In order to prevent bias in the data evaluation process, each baby will be numbered by the researcher during the application and these numbers will be used by the statistical expert in statistical evaluations. The statistical expert will not learn the identity information of the participants and will only perform statistics according to the numbering.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foot massage group (Experimental): Foot massage will be performed by the researcher for 10 minutes on two consecutive days a week in the infants' own homes. In foot massage, euphlorage, petrisage and friction techniques will be used in the appropriate order.
  Infants in the foot massage group will be visited five times in total, two times each in the first encounter, first and second weeks. Related forms (Infantile colic and newborn comfort behavior scale) will be filled out by the researcher three times in total, once for the first encounter and once for each week. A total of two forms related to crying and sleep, one for each week, will be completed by the mother at the end of the study. The maternal state-trait anxiety scale will be completed twice, at the first encounter and at the end of the intervention.
  Interventions: Other: Foot massage
- Mother heart sound group (Experimental): For the group to listen to the mother's heart sounds, the heart sounds of the mothers of the babies will be recorded on an mp3 player in a quiet environment (in their own homes) with the help of hand-held doopes. The volume (65 decibels) and distance of the mp3 player will be determined by the researcher with the help of a decibel meter and the appropriate distance will be determined. The mother will play this sound to the infant for half an hour every day for two weeks, in coordination with the hours of the intervention in the other groups.
  The infants in this group will be visited three times in total, once at the first encounter and once at the end of the first and second weekends, and the relevant forms (Infantile colic and newborn comfort behavior, state-trait anxiety scale) will be applied. Forms related to crying and sleep will be completed by the mother two times in total, one for each week.
  Interventions: Other: Mother heart sound
- Foot massage and mother heart sound group (mixed group) (Experimental): For the group in which maternal heart sounds and foot massage will be applied, the heart sounds of the mothers of the babies will be recorded on an mp3 player in a quiet environment (in their own homes) with the help of hand-held doopes. The sound (65 decibels) and distance of the mp3 player will be determined by the researcher with the help of a decibel meter. The researcher will perform foot massage as in the massage group and the mother's heart sound will be played for a total of half an hour with the massage. The infants in this group will be visited five times in total, once in the first encounter and twice each in the first and second week, and the relevant forms (Infantile colic, neonatal comfort behavior scales will be applied 3 times for infants; state-trait anxiety scale will be applied twice for the mother, once at the beginning and twice at the end). A total of two forms related to crying and sleep will be completed by the mother, one for each week.
  Interventions: Other: Foot massage and maternal heart sound

INTERVENTIONS:
Other: Foot massage — Infants in the foot massage group will receive foot massage by the researcher on two consecutive days of the week for a total of four times. The massage will be performed in accordance with the specified application steps for 10 minutes just before the baby's restlessness starts.
  Arms: Foot massage group
Other: Mother heart sound — The sound recorded by the researcher under appropriate conditions will be played to the babies in the maternal heart sound group from an appropriate distance. The sound will be played a total of four times, on two consecutive days of the week, just before the baby's restlessness begins and for half an hour.
  Arms: Mother heart sound group
Other: Foot massage and maternal heart sound — Infants in the foot massage and maternal heart sound group will receive foot massage by the researcher on two consecutive days of the week for a total of four times. The massage will be performed in accordance with the specified application steps for 10 minutes just before the baby's restlessness starts. From the beginning of the massage, the pre-recorded maternal heart sound will be played to the infant for 30 minutes from an appropriate distance.
  Arms: Foot massage and mother heart sound group (mixed group)

SUMMARY:
Infantile colic is a developmental disorder that reduces comfort levels in infants with intense crying crises and has negative effects on the infant and family. The study is planned to measure the effect of the combination of maternal heart sound simulation, aromatic foot massage and maternal heart sound simulation and aromatic foot massage on the colic and comfort levels of infants with infantile colic. It is aimed to alleviate colic symptoms, increase comfort levels, regulate daily crying and sleep durations (increase in sleep durations, decrease in crying durations) and support the development of infants in this context by using maternal heart sound simulation, aromatic foot massage and their combined application.

DETAILED DESCRIPTION:
Infantile colic is a developmental disorder that occurs in the second week of extrauterine life, reaches its peak in the sixth week, continues up to four to six months, and negatively affects the infant and family in healthy infants who develop rapidly. Infantile colic is a very common disorder among functional gastrointestinal diseases. When the studies conducted to determine the prevalence of infantile colic are examined, it is seen that the prevalence varies according to the development level of the countries (prevalence increases as the development level decreases) and the average figures are %5-25.

Although there are many studies on infantile colic, there is no clear acceptance about its etiology. Regarding the etiology of infantile colic; it is mentioned that gastrointestinal, psychosocial and immature central nervous system causes may be triggering in the disease. In addition, low birth weight, lactose intolerance, food allergy (cow's milk), hypersensitivity, excessive gas, increased peristalsis, bottle feeding, swallowing excess air during crying, gastroesophageal reflux, perception of distension as pain due to immature intestinal structure, incompatibility in serotonin and melatonin circadian rhythm in the first three months, as well as factors such as family stress, anxiety and psychosocial problems in the mother may play a role in the disease.

In functional gastrointestinal disorders, the lack of a structural, anatomical or biochemical impairment that can provide an objective assessment of the disease makes the diagnostic process difficult. Considering the lack of verbal expression in infants, it is essential to use certain accepted criteria in the diagnostic process in order to make an objective diagnosis of the disease. Due to these requirements, the Wessel technique and Rome II-III-IV criteria were used in the diagnostic process of infantile colic, respectively, and the use of Wessel, Rome III-IV is still ongoing. The first description of infantile colic in infants was made by Wessel (1954). Wessel defined infantile colic as crying for more than three hours a day, for more than three days a week and for more than three weeks without any developmental or situational discomfort. The first use of a child-specific FGID diagnosis was in the Rome II criteria in 1999. The use of Rome II criteria did not meet the need due to lack of literature and evidence. Therefore, with the publication of Rome III criteria in 2006, the diagnostic process became more objective. With the studies conducted over the years, Rome III diagnostic criteria were revised in 2006 and Rome IV diagnostic criteria were started to be used in order to better understand the diseases and provide the best treatment.

Although there is no fixed treatment protocol in the treatment of infantile colic, pharmacological and non-pharmacological methods are used. Although pharmacological agents are occasionally used in treatment, dietary and behavioral treatment methods are mostly used in the treatment of the disease. Although pharmacologic treatment is occasionally used in infantile colic, studies do not support the use of any pharmacologic agent within the scope of evidence-based practice. In the pharmacologic treatment of infantile colic; Although drug groups such as anelgesics, antispasmolytics (especially simethicone, dicyclomine) and proton pump inhibitors are used, there is no evidence-based practice with usability because there is no specific treatment.

Since the foods consumed by the mother may affect the baby through milk, it is recommended to temporarily exclude foods such as citrus fruits, eggs, cola, cow's milk, chocolate, dried legumes, nuts and dairy products from the mother's diet. Herbal teas may improve the symptoms of infantile colic and may also provide sedation, but caution should be exercised because the level of evidence is not sufficient. The use of probiotics is another method that may alleviate colic symptoms because it improves the intestinal microbiota, and the use of hydrolyzed formulas with prebiotics is recommended in infants fed formula.

In most FGIDs such as infantile colic, supportive therapies, therapeutic communication and approach techniques are prioritized. In FGIDs in infants, direct behavioral therapy methods are frequently used among non-pharmacological treatments and positive effects are reported. Direct behavioral therapy methods include sensorimotor stimulation (auditory stimuli, therapeutic touch, etc.), therapeutic massage, reflexology, not exposing the baby to excessive stimuli, rocking the baby or moving the baby in a car, kangaroo, etc. (kangaroo care), using a pacifier, applying warmth to the abdomen, swaddling the baby in a way that does not squeeze the baby, and warm baths. In addition to direct behavioral therapy methods, practices such as dietary changes, nutritional recommendations, glucose-sucrose applications, probiotic and herbal supplements, acupuncture and spinal manipulation to reduce the frequency and severity of infantile colic symptoms are also used in non-pharmacological treatment.

Massage is the art of touch that concerns all or part of the body and creates a relaxing effect in the area where it is applied. Massage practice in infants also positively affects the baby's attachment process due to health, comfort of life and sensual contact. Massage application is an application that supports the coordination process with muscle stimulation and has positive effects on physical development, circulatory, respiratory and digestive systems. Massage, whose positive effects on colic symptoms are frequently emphasized in studies, also contributes to sleep duration as it also provides relaxation for the baby.

Techniques such as euphlorage, petrissage, friction, vibration and percussion are used in massage application. In baby foot massage applications, euphlorage, petrissage and friction techniques are frequently preferred. Öfloraj; It is a patting movement applied towards the direction of venous circulation returning to the heart, which stimulates nerve, blood and lymph circulation, sweat and sebaceous glands by affecting the skin and subcutaneous tissues. Petrisage is a kneading movement applied by taking the subcutaneous tissue and muscles between the thumb and other fingers. It increases the circulation of the muscles and ensures the removal of metabolic waste products. Friction is a sliding and pressing movement applied to the body surface in small circles with fingertips in order to loosen the fluid accumulations in the skin and subcutaneous tissues with lymph circulation and stiffness around the joints.

Comfort is defined as the individual being comfortable, reducing stress and painful situations and making life easier. Comfort in newborns and infants includes indicators whose forms of expression differ from those of adults and are important in maintaining healthy development. Comfort indicators in newborns; Pulse and respiratory rate within normal limits and regularity Minimal body color changes Order in body movements Active use of behaviors that relax the newborn A healthy growth and development process It is defined as the realization of discharge as soon as possible. It is important for the sustainability of growth and development that babies are exposed to less pain and stress at birth. The pain experienced by babies in infantile colic creates distress for them and reduces the comfort level in both the baby and the family. Nursing is a special occupational group in which complementary, care-oriented practices are frequently used, based on holistic care philosophy, and caring about the support and sustainability of health. Nurses are the professionals who will perform these practices in complementary treatment. Nursing care applied systematically in infantile colic contributes to the health of the baby and family. A good family support programming, education, counseling, strengthening support factors and ensuring effective practices, implemented by taking all variables into consideration, will reduce the symptoms of infantile colic, while at the same time supporting infant and family attachment, spending more quality time and strengthening family ties, while reducing the frequency or severity of negative experiences that family members experience / may experience such as inadequacy and helplessness. Thus, family members will be helped to prevent/reduce psychological problems that may be seen due to infantile colic and the comfort of life will increase for both the baby and the family.

ELIGIBILITY:
Inclusion criteria:

* Babies crying more than three hours a day, three days a week, according to the Wessel technique,
* Babies are between 2 and 16 weeks postpartum,
* The baby does not have any other illness that may cause restlessness and crying,
* The baby does not have a chronic disease,
* Absence of any anomaly in the foot area that would prevent massage,
* Babies have passed the hearing test,
* Babies do not have a problem that prevents hearing,
* Infants are not receiving pharmacologic treatment for infantile colic,
* Infants are not receiving non-pharmacologic treatment for infantile colic,
* Babies are not receiving any pharmacologic (analgesic/sedative) treatment that may affect pain and comfort.

Exclusion and exclusion criteria:

* Initiation of any pharmacologic treatment that may affect colic, comfort, sleep and crying times in infants included in the study,
* Initiation of any non-pharmacologic treatment that may affect colic, comfort, sleep and crying times in infants included in the study,
* Incomplete data.

Ages: 2 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in colic scale ratings induced by maternal heart sound | Two weeks
  The colic scale consists of 19 questions. The minimum score that can be obtained from the scale in total is 19 and the maximum score is 114. A score of 48 and above on the scale indicates the presence of colic.After 48 points, each point increase indicates an increase in the severity of colic
Changes in comfort scale ratings as a result of maternal heart sound | Two weeks
  The comfort scale consists of 6 sub-dimensions.Each sub-dimension is evaluated between 1 and 5 points. Comfort is considered good if the total score is 15 or above, and inadequate if it is below.
Changes in colic scale assessments induced by foot massage | Two weeks
  The colic scale consists of 19 questions. The minimum score that can be obtained from the scale in total is 19 and the maximum score is 114. A score of 48 and above on the scale indicates the presence of colic.After 48 points, each point increase indicates an increase in the severity of colic
Changes in comfort scale assessments induced by foot massage | Two weeks
  The comfort scale consists of 6 sub-dimensions.Each sub-dimension is evaluated between 1 and 5 points. Comfort is considered good if the total score is 15 or above, and inadequate if it is below.

CONTACTS AND LOCATIONS:
Overall Officials: Nejla CANBULAT ŞAHİNER, Professor, Study Director — Karamanoğlu Mehmetbey University Faculty of Health Sciences
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study is a doctoral thesis and the data collection process is ongoing. For this reason, it is planned to share only the title until the study is finalized and the whole study at the end of the study.

REFERENCES:
- [Background] Aagaard K, Ma J, Antony KM, Ganu R, Petrosino J, Versalovic J. The placenta harbors a unique microbiome. Sci Transl Med. 2014 May 21;6(237):237ra65. doi: 10.1126/scitranslmed.3008599. PMID 24848255
- [Background] Ahmed M, Billoo AG, Iqbal K, Memon A. Clinical Efficacy Of Lactase Enzyme Supplement In Infant Colic: A Randomised Controlled Trial. J Pak Med Assoc. 2018 Dec;68(12):1744-1747. PMID 30504935
- [Background] Baldassarre ME, Di Mauro A, Mastromarino P, Fanelli M, Martinelli D, Urbano F, Capobianco D, Laforgia N. Administration of a Multi-Strain Probiotic Product to Women in the Perinatal Period Differentially Affects the Breast Milk Cytokine Profile and May Have Beneficial Effects on Neonatal Gastrointestinal Functional Symptoms. A Randomized Clinical Trial. Nutrients. 2016 Oct 27;8(11):677. doi: 10.3390/nu8110677. PMID 27801789
- [Background] Bellaiche M, Ategbo S, Krumholz F, Ludwig T, Miqdady M, Abkari A, Vandenplas Y. A large-scale study to describe the prevalence, characteristics and management of functional gastrointestinal disorders in African infants. Acta Paediatr. 2020 Nov;109(11):2366-2373. doi: 10.1111/apa.15248. Epub 2020 Mar 18. PMID 32150302
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Background] Chogle A, Velasco-Benitez CA, Koppen IJ, Moreno JE, Ramirez Hernandez CR, Saps M. A Population-Based Study on the Epidemiology of Functional Gastrointestinal Disorders in Young Children. J Pediatr. 2016 Dec;179:139-143.e1. doi: 10.1016/j.jpeds.2016.08.095. Epub 2016 Oct 7. PMID 27726867
- [Background] Coughlin M, Gibbins S, Hoath S. Core measures for developmentally supportive care in neonatal intensive care units: theory, precedence and practice. J Adv Nurs. 2009 Oct;65(10):2239-48. doi: 10.1111/j.1365-2648.2009.05052.x. PMID 19686402
- [Background] Çelik, H.İ., Elbasan, B., Gücüyener, K., Kayıhan, H. ve Huri, M., Investigation of Sensory Processing Skills in Preterm and Term Infants. Physiotherapy Rehabilitation, 2018; 29 (2): 31-36. doi: 10.21653/tjpr.343255.
- [Background] Cetinkaya B, Basbakkal Z. A validity and reliability study investigating the Turkish version of the Infant Colic Scale. Gastroenterol Nurs. 2007 Mar-Apr;30(2):84-90; discussion 90. doi: 10.1097/01.SGA.0000267925.31803.30. PMID 17440307
- [Background] Cetinkaya B, Basbakkal Z. The effectiveness of aromatherapy massage using lavender oil as a treatment for infantile colic. Int J Nurs Pract. 2012 Apr;18(2):164-9. doi: 10.1111/j.1440-172X.2012.02015.x. PMID 22435980
- [Background] Dos Reis Buzzo Zermiani AP, de Paula Soares ALPP, da Silva Guedes de Moura BL, Miguel ERA, Lopes LDG, de Carvalho Scharf Santana N, da Silva Santos T, Demarchi IG, Teixeira JJ. Evidence of Lactobacillus reuteri to reduce colic in breastfed babies: Systematic review and meta-analysis. Complement Ther Med. 2021 Dec;63:102781. doi: 10.1016/j.ctim.2021.102781. Epub 2021 Oct 7. PMID 34627993
- [Background] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Background] Cirgin Ellett ML, Murphy D, Stroud L, Shelton RA, Sullivan A, Ellett SG, Ellett LD. Development and psychometric testing of the infant colic scale. Gastroenterol Nurs. 2003 May-Jun;26(3):96-103. doi: 10.1097/00001610-200305000-00002. PMID 12811319
- [Background] Gelfand AA, Thomas KC, Goadsby PJ. Before the headache: infant colic as an early life expression of migraine. Neurology. 2012 Sep 25;79(13):1392-6. doi: 10.1212/WNL.0b013e31826c1b7b. Epub 2012 Sep 12. PMID 22972642
- [Background] Gordon M, Gohil J, Banks SS. Parent training programmes for managing infantile colic. Cochrane Database Syst Rev. 2019 Dec 3;12(12):CD012459. doi: 10.1002/14651858.CD012459.pub2. PMID 31794639
- [Background] Hill DJ, Roy N, Heine RG, Hosking CS, Francis DE, Brown J, Speirs B, Sadowsky J, Carlin JB. Effect of a low-allergen maternal diet on colic among breastfed infants: a randomized, controlled trial. Pediatrics. 2005 Nov;116(5):e709-15. doi: 10.1542/peds.2005-0147. PMID 16263986
- [Background] Johnson JD, Cocker K, Chang E. Infantile Colic: Recognition and Treatment. Am Fam Physician. 2015 Oct 1;92(7):577-82. PMID 26447441
- [Background] Johnson JM, Adams ED. The Gastrointestinal Microbiome in Infant Colic: A Scoping Review. MCN Am J Matern Child Nurs. 2022 Jul-Aug 01;47(4):195-206. doi: 10.1097/NMC.0000000000000832. PMID 35352686
- [Background] Kahraman, A., Başbakkal, Z. ve Yalaz, M., Validity and Reliability of the Newborn Comfort Behavior Scale. Journal of Nursing Research. 2014; 1: 1-11.
- [Background] Kanbir, O., Classical Massage, Treatment, Sports Massage, Classical Massage Rest, Ekin Publishing, 5th Edition, Bursa, 2015; 135-157.
- [Background] Karakoc A, Turker F. Effects of white noise and holding on pain perception in newborns. Pain Manag Nurs. 2014 Dec;15(4):864-70. doi: 10.1016/j.pmn.2014.01.002. Epub 2014 Feb 20. PMID 24559599
- [Background] Keefe MR, Kajrlsen KA, Lobo ML, Kotzer AM, Dudley WN. Reducing parenting stress in families with irritable infants. Nurs Res. 2006 May-Jun;55(3):198-205. doi: 10.1097/00006199-200605000-00006. PMID 16708044
- [Background] Koppen IJ, Nurko S, Saps M, Di Lorenzo C, Benninga MA. The pediatric Rome IV criteria: what's new? Expert Rev Gastroenterol Hepatol. 2017 Mar;11(3):193-201. doi: 10.1080/17474124.2017.1282820. Epub 2017 Jan 24. PMID 28092724
- [Background] Korpela K, Renko M, Paalanne N, Vanni P, Salo J, Tejesvi M, Koivusaari P, Pokka T, Kaukola T, Pirttila AM, Tapiainen T. Microbiome of the first stool after birth and infantile colic. Pediatr Res. 2020 Nov;88(5):776-783. doi: 10.1038/s41390-020-0804-y. Epub 2020 Feb 13. PMID 32053826
- [Background] Mai T, Fatheree NY, Gleason W, Liu Y, Rhoads JM. Infantile Colic: New Insights into an Old Problem. Gastroenterol Clin North Am. 2018 Dec;47(4):829-844. doi: 10.1016/j.gtc.2018.07.008. Epub 2018 Sep 28. PMID 30337035
- [Background] McKenzie SA. Fifteen-minute consultation: Troublesome crying in infancy. Arch Dis Child Educ Pract Ed. 2013 Dec;98(6):209-11. doi: 10.1136/archdischild-2013-303903. Epub 2013 Aug 26. PMID 23979927
- [Background] Narang M, Shah D. Oral lactase for infantile colic: a randomized double-blind placebo-controlled trial. BMC Pediatr. 2022 Aug 3;22(1):468. doi: 10.1186/s12887-022-03531-8. PMID 35922776
- [Background] Obermayr F, Seitz G. Recent developments in cell-based ENS regeneration - a short review. Innov Surg Sci. 2018 Mar 9;3(2):93-99. doi: 10.1515/iss-2018-0005. eCollection 2018 Jun. PMID 31579772
- [Background] Perry R, Leach V, Penfold C, Davies P. An overview of systematic reviews of complementary and alternative therapies for infantile colic. Syst Rev. 2019 Nov 11;8(1):271. doi: 10.1186/s13643-019-1191-5. PMID 31711532
- [Background] Sarasu JM, Narang M, Shah D. Infantile Colic: An Update. Indian Pediatr. 2018 Nov 15;55(11):979-987. Epub 2018 Jun 13. PMID 29941700
- [Background] Savino F, Quartieri A, De Marco A, Garro M, Amaretti A, Raimondi S, Simone M, Rossi M. Comparison of formula-fed infants with and without colic revealed significant differences in total bacteria, Enterobacteriaceae and faecal ammonia. Acta Paediatr. 2017 Apr;106(4):573-578. doi: 10.1111/apa.13642. Epub 2016 Nov 15. PMID 27763733
- [Background] Savino F, Garro M, Montanari P, Galliano I, Bergallo M. Crying Time and RORgamma/FOXP3 Expression in Lactobacillus reuteri DSM17938-Treated Infants with Colic: A Randomized Trial. J Pediatr. 2018 Jan;192:171-177.e1. doi: 10.1016/j.jpeds.2017.08.062. Epub 2017 Sep 29. PMID 28969887
- [Background] Steutel NF, Zeevenhooven J, Scarpato E, Vandenplas Y, Tabbers MM, Staiano A, Benninga MA. Prevalence of Functional Gastrointestinal Disorders in European Infants and Toddlers. J Pediatr. 2020 Jun;221:107-114. doi: 10.1016/j.jpeds.2020.02.076. PMID 32446468
- [Background] Schreck Bird A, Gregory PJ, Jalloh MA, Risoldi Cochrane Z, Hein DJ. Probiotics for the Treatment of Infantile Colic: A Systematic Review. J Pharm Pract. 2017 Jun;30(3):366-374. doi: 10.1177/0897190016634516. Epub 2016 Mar 2. PMID 26940647
- [Background] Shirazinia R, Golabchifar AA, Fazeli MR. Efficacy of probiotics for managing infantile colic due to their anti-inflammatory properties: a meta-analysis and systematic review. Clin Exp Pediatr. 2021 Dec;64(12):642-651. doi: 10.3345/cep.2020.01676. Epub 2021 Apr 12. PMID 33848417
- [Background] Wolke D, Bilgin A, Samara M. Systematic Review and Meta-Analysis: Fussing and Crying Durations and Prevalence of Colic in Infants. J Pediatr. 2017 Jun;185:55-61.e4. doi: 10.1016/j.jpeds.2017.02.020. Epub 2017 Apr 3. PMID 28385295
- [Background] de Weerth C, Fuentes S, Puylaert P, de Vos WM. Intestinal microbiota of infants with colic: development and specific signatures. Pediatrics. 2013 Feb;131(2):e550-8. doi: 10.1542/peds.2012-1449. Epub 2013 Jan 14. PMID 23319531
- [Background] de Weerth C, Fuentes S, de Vos WM. Crying in infants: on the possible role of intestinal microbiota in the development of colic. Gut Microbes. 2013 Sep-Oct;4(5):416-21. doi: 10.4161/gmic.26041. Epub 2013 Aug 9. PMID 23941920
- [Background] Yavaş, Çelik, M., Comparison of White Noise and Massage Application Methods in 0-12 Month Colicky Infants. Master's Thesis, Çukurova University Institute of Health Sciences, Adana. 2015.
- [Background] Yavaş, Çelik, M. Infantile Colic and Nursing Approaches. Turkey Clinics, 2016; 8 (4), 335-342.
- [Background] Iacovou M, Ralston RA, Muir J, Walker KZ, Truby H. Dietary management of infantile colic: a systematic review. Matern Child Health J. 2012 Aug;16(6):1319-31. doi: 10.1007/s10995-011-0842-5. PMID 21710185
- [Background] Zeevenhooven J, Koppen IJ, Benninga MA. The New Rome IV Criteria for Functional Gastrointestinal Disorders in Infants and Toddlers. Pediatr Gastroenterol Hepatol Nutr. 2017 Mar;20(1):1-13. doi: 10.5223/pghn.2017.20.1.1. Epub 2017 Mar 27. PMID 28401050
- [Background] Zeevenhooven J, Browne PD, L'Hoir MP, de Weerth C, Benninga MA. Infant colic: mechanisms and management. Nat Rev Gastroenterol Hepatol. 2018 Aug;15(8):479-496. doi: 10.1038/s41575-018-0008-7. PMID 29760502
- See also: Alves, J.G.B., De Brito, R.C.C.M. ve Cavalcanti, T.S., (2012). Effectiveness of Mentha piperita in the Treatment of Infantile Colic: A Crossover Study. Evid Based Complement Alternat Med., 981352. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3403674/
- See also: Roma vakfı — http://theromefoundation.org/rome-iv/rome-iv-criteria/
- See also: Roma vakfı — http://theromefoundation.org/rome-iv/whats-new-for-rome-iv/
- See also: Yıldız, S. ve Coşkun, P., (2023). Doğal ve Yapay Tatlandırıcıların Sağlık Açısından İncelenmesi. Sağlık Bilimlerinde Yenilikçi Çalışmalar, 775-791. (Online Kitap Bölümü, 41. bölüm — https://scholar.google.com.tr/scholar?q=Do%C4%9Fal+ve+Yapay+Tatland%C4%B1r%C4%B1c%C4%B1lar%C4%B1n+Sa%C4%9Fl%C4%B1k+A%C3%A7%C4%B1s%C4%B1ndan+%C4%B0ncelenmesi&hl=tr&as_sdt=0&as_vis=1&oi=scholart